CLINICAL TRIAL: NCT02028767
Title: Bioequivalence of Empagliflozin/Metformin (12.5mg/500mg) Fixed Dose Combination Tablets Compared to Tablets Administered Together in Healthy Male and Female Volunteers Under Fed Conditions (an Open Label, Randomised, Single Dose, Two Period, Two Sequence Crossover Study)
Brief Title: Bioequivalence Study in Healthy Volunteers for Empagliflozin/Metformin Fixed Dose Combination Compared to Separate Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1276.24
Record Dates: First submitted 2014-01-06; First posted 2014-01-07 (Estimated); Results first posted 2015-07-24 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-06

CONDITIONS: Healthy
MeSH Terms: interventions — empagliflozin; Metformin

ARMS (2):
- Fixed Dose Combination (FDC) (Experimental): 12.5 mg Empagliflozin / 500mg metformin fixed dose combination
  Interventions: Drug: Empagliflozin/Metformin FDC
- Separate tablets (Active Comparator): Empagliflozin and Metformin tablets
  Interventions: Drug: Empagliflozin 2.5 mg; Drug: Empagliflozin 10 mg; Drug: Metformin 500 mg

INTERVENTIONS:
Drug: Empagliflozin 2.5 mg — Empagliflozin 2.5 mg tablet
  Arms: Separate tablets
Drug: Empagliflozin 10 mg — Empagliflozin 10 mg tablet
  Arms: Separate tablets
Drug: Metformin 500 mg — Metformin 500 mg tablet
  Arms: Separate tablets
Drug: Empagliflozin/Metformin FDC — 12.5 mg Empagliflozin / 500 mg Metformin
  Arms: Fixed Dose Combination (FDC)

SUMMARY:
The trial is being conducted to establish the bioequivalence of emp/met (12.5mg/500mg) fixed dose combination tablets compared to tablets administered together in healthy male and female volunteers under fed conditions.

ELIGIBILITY:
Inclusion criteria:

1. Healthy males or females according to the investigator's assessment, as based on the following criteria: a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG and clinical laboratory tests.
2. Age 18 to 50 years (inclusive)
3. BMI 18.5 to 29.9 kg/m2 (inclusive)
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation.

Exclusion criteria:

1. Any finding in the medical examination (Including blood pressure [BP], pulse rate [PR], or electrocardiogram [ECG]) deviating from normal and judged clinically relevant by the investigator.
2. Any evidence of a concomitant disease judged clinically relevant by the investigator.
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders.
4. Surgery of the gastrointestinal tract that could interfere with kinetics of the study drug(s)
5. Diseases of the central nervous system (such as epilepsy), other neurological disorders or psychiatric disorders.
6. History of relevant orthostatic hypotension, fainting spells, or blackouts.
7. Chronic or relevant acute infections
8. History of relevant allergy/hypersensitivity (including allergy to the trial medication or it's excipients)
9. Intake of drugs with a long half-life (>24 hours) within 30 days or less than 10 half-lives of the respective drug prior to administration of trial medication.
10. Within 14 days prior to the administration of trial medication, use of drugs that might reasonably influence the results of the trial, based on current knowledge
11. Participation in another trial with investigational drug administration within 60 days prior to administration of trial medication.
12. Smoker (has used tobacco or nicotine-containing products within 6 months prior to administration of trial medication)
13. Inability to refrain from smoking on specified trial days
14. Alcohol abuse (consumption of more than 20g/day in females and 30g/day in males or > 7 alcohol-containing drinks per week)
15. Drug abuse or positive drug screen
16. Blood donation (more than 100 ml wihtin 30 days prior to administration of trial medication or intended during the trial)
17. Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
18. Inability to comply with dietary regimen of trial site
19. Subject is assessed by the investigator as unsuitable for inclusion, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study.

    For female subjects:
20. Positive pregnancy test, pregnancy or plans to become pregnant within 30 days after study completion.
21. No adequate contraception during the study and until 1 month after study completion, i.e. not any of the following: implants, injectables, combined oral contraceptives, IUD (intrauterine device), sexual abstinence for at least 1 month prior to enrolment, vasectomised partner (vasectomy performed at least 1 year prior to enrolment), or surgical sterilisation (including hysterectomy). Females, who do not have a vasectomised partner, are not sexually abstinent, surgically sterile, or post menopausal will be asked to use an additional barrier method (e.g. condom, diaphragm with spermicide). Post-menopausal is defined as at least 1 year of spontaneous amenorrhea and deemed post menopausal by a physician based on screening clinical laboratory tests (follicle stimulating hormone and luteinizing hormone).
22. Lactation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1276.24.001 Boehringer Ingelheim Investigational Site, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Fixed Dose Combination (FDC) First, Then Separate Tablets: Empagliflozin / Metformin FDC: 12.5 mg Empagliflozin / 500 mg Metformin first,
  then free combination of Empagliflozin 2.5 mg tablet, Empagliflozin 10 mg tablet and Metformin 500 mg tablet
  Both medications were administered oral with 240 mL water after intake of a high-fat, high-calorie meal.
- Separate Tablets First, Then Fixed Dose Combination (FDC): free combination of Empagliflozin 2.5 mg tablet, Empagliflozin 10 mg tablet and Metformin 500 mg tablet first,
  then Empagliflozin / Metformin FDC: 12.5 mg Empagliflozin / 500 mg Metformin
  Both medications were administered oral with 240 mL water after intake of a high-fat, high-calorie meal.
Period: Treatment Period 1
Arm/Group | Fixed Dose Combination (FDC) First, Then Separate Tablets | Separate Tablets First, Then Fixed Dose Combination (FDC)
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0
Period: Treatment Period 2
Arm/Group | Fixed Dose Combination (FDC) First, Then Separate Tablets | Separate Tablets First, Then Fixed Dose Combination (FDC)
Started | 16 | 16
Completed | 14 | 16
Not Completed | 2 | 0
Not completed — Non compliant with protocol | 1 | 0
Not completed — Reason other than those specified above | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): includes all subjects who were dispensed study medication and were documented to have received at least 1 dose of study medication.
Groups:
- Fixed Dose Combination vs. Separate Tablets: 12.5 mg Empagliflozin / 500mg metformin fixed dose combination vs. free combination of 2.5 mg tablet Empagliflozin, 10 mg tablet Empagliflozin and 500 mg tablet Metformin
Arm/Group | Fixed Dose Combination vs. Separate Tablets
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: AUC (0-tz) (Area Under the Concentration-time Curve of Metformin in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point)
Description: AUC (0-tz) (area under the concentration-time curve of metformin in plasma over the time interval from 0 to the last quantifiable data point)
Time Frame: 1 hour (h) before drug administration and 20 minutes (min), 40min, 1h, 1h 30min, 2h, 2h 30min, 3h, 3h 30min, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 34h, 48h and 72h after drug administration
Population: Pharmacokinetic set (PKS): includes all subjects of the TS who provided at least 1 observation for at least 1 primary pharmacokinetic endpoint, and had no important protocol violations with respect to the statistical evaluation of pharmacokinetic endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Fixed Dose Combination (FDC): 12.5 mg Empagliflozin / 500mg metformin fixed dose combination
  Empagliflozin / Metformin FDC: 12.5 mg Empagliflozin / 500 mg Metformin
Arm/Group | Fixed Dose Combination (FDC) | Separate Tablets
Number analyzed (Participants) | 32 | 30
ng*h/mL | 6260 (20.4) | 6360 (21.8)
Statistical Analysis 1: Comparison: Fixed Dose Combination (FDC) vs Separate Tablets; Test type: Non-Inferiority or Equivalence — Bioequivalence test; p = 0.0000, ANOVA — The p-value relates to the null hypothesis of non-equivalence; Geometric mean ratio = 98.57, 90% CI 2-sided [94.662 to 102.639], Standard Error of Mean 1.024 — The geometric mean ratio is the exponential of the estimated mean difference on the log-scale between 'FDC' and 'Separate tablets'. ANOVA on the log scale: sequence, period and treatment as fixed effects; subjects within sequences as random effect
Statistical Analysis 2: Comparison: Fixed Dose Combination (FDC) vs Separate Tablets; Analysis with fixed effects for all terms; Test type: Non-Inferiority or Equivalence — Bioequivalence test; p < 0.0001, ANOVA — The p-value relates to the null hypothesis of non-equivalence; Geometric mean ratio = 98.71, 90% CI 2-sided [94.783 to 102.796], Standard Error of Mean 1.024 — The geometric mean ratio is the exponential of the estimated mean difference on the log-scale between 'FDC' and 'Separate tablets'. ANOVA on the log-scale: sequence, subjects within sequences, period and treatment as fixed effects

2. Primary Outcome: Cmax (Maximum Measured Concentration of Metformin in Plasma)
Description: Cmax (maximum measured concentration of metformin in plasma)
Time Frame: as for outcome 1
Population: PKS: includes all subjects of the TS who provided at least 1 observation for at least 1 primary pharmacokinetic endpoint, and had no important protocol violations with respect to the statistical evaluation of pharmacokinetic endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Fixed Dose Combination (FDC) | Separate Tablets
Number analyzed (Participants) | 32 | 30
ng/mL | 746 (21.3) | 754 (23.3)
Statistical Analysis 1: Comparison: Fixed Dose Combination (FDC) vs Separate Tablets; Test type: Non-Inferiority or Equivalence — Bioequivalence test; p = 0.0000, ANOVA — The p-value relates to the null hypothesis of non-equivalence; Geometric mean ratio = 98.93, 90% CI 2-sided [95.856 to 102.107], Standard Error of Mean 1.019 — The geometric mean ratio is the exponential of the estimated mean difference on the log-scale between 'FDC' and 'Separate tablets'. ANOVA on the log-scale: sequence, period and treatment as fixed effects; subjects within sequences as random effect
Statistical Analysis 2: Comparison: Fixed Dose Combination (FDC) vs Separate Tablets; Analysis with fixed effects for all terms; Test type: Non-Inferiority or Equivalence — Bioequivalence test; p < 0.0001, ANOVA — The p-value relates to the null hypothesis of non-equivalence; Geometric mean ratio = 98.96, 90% CI 2-sided [95.877 to 102.150], Standard Error of Mean 1.019 — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: AUC (0-infinity) (Area Under the Concentration-time Curve of Metformin in Plasma Over the Time Interval From 0 Extrapolated to Infinity)
Description: AUC (0-infinity) (Area under the concentration-time curve of metformin in plasma over the time interval from 0 extrapolated to infinity)
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Fixed Dose Combination (FDC) | Separate Tablets
Number analyzed (Participants) | 32 | 30
ng*h/mL | 6410 (20.9) | 6520 (22.5)
Statistical Analysis 1: Comparison: Fixed Dose Combination (FDC) vs Separate Tablets; Test type: Non-Inferiority or Equivalence — Bioequivalence test; p = 0.0000, ANOVA — The p-value relates to the null hypothesis of non-equivalence; Geometric mean ratio = 98.28, 90% CI 2-sided [94.549 to 102.156], Standard Error of Mean 1.023 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Fixed Dose Combination (FDC) vs Separate Tablets; Analysis with fixed effects for all terms; Test type: Non-Inferiority or Equivalence — Bioequivalence test; p < 0.0001, ANOVA; The p-value relates to the null hypothesis of non-equivalence; Geometric mean ratio = 98.35, 90% CI 2-sided [94.603 to 102.252], Standard Error of Mean 1.023 — [estimate comment as in outcome 1, analysis 2]

ADVERSE EVENTS:
Time Frame: From first trial medication intake until next intake or the day after the end-of-trial visit, 16 days
Arm/Group | Fixed Dose Combination (FDC) | Separate Tablets
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/30
Other Adverse Events (participants affected / at risk) | 11/32 | 5/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fixed Dose Combination (FDC) (N=32) | Separate Tablets (N=30)
Somnolence (Nervous system disorders) | 7 | 4
Headache (Nervous system disorders) | 4 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.